CLINICAL TRIAL: NCT03279081
Title: A Phase-III, Randomized, Double-blind, Parallel-group, Placebo-controlled, International, Multicentre Study to Assess Efficacy and Safety of Cx601, Adult Allogeneic Expanded Adipose-derived Stem Cells (eASC) for the Treatment of Complex Perianal Fistula(s) in Patients With Crohn's Disease Over a Period of 24 Weeks and a Follow-up Period up to 52 Weeks
Brief Title: Study to Assess Efficacy and Safety of Cx601, Adult Allogeneic Expanded Adipose-derived Stem Cells (eASC) for the Treatment of Complex Perianal Fistula(s) in Participants With Crohn's Disease (CD)
Acronym: ADMIRE-CD-II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tigenix S.A.U. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cx601-0303; 2017-000725-12 (EudraCT Number)
Record Dates: First submitted 2017-07-21; First posted 2017-09-12 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; complex perianal fistula(s)
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (saline) 24 milliliters (mL) was administered once by local injection.
  Interventions: Other: Placebo
- Cx601 (Experimental): Cx601 expanded adipose-derived stem cells (eASCs) 120 million cells (5 million cells per mL) was administered once by local injection.
  Interventions: Drug: Cx601

INTERVENTIONS:
Drug: Cx601 — Cx601 eASCs intralesional injection.
  Arms: Cx601
Other: Placebo — Cx601 placebo-matching eASCs intralesional injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the combined remission of complex perianal fistulas, defined as the clinical assessment at Week 24 of closure of all treated external openings that were draining at baseline despite gentle finger compression, and absence of collections greater than (>) 2 centimeter (cm) (in at least 2 dimensions) confirmed by blinded central magnetic resonance imaging (MRI) assessment at Week 24.

DETAILED DESCRIPTION:
This study is to assess the efficacy and safety of Cx601, eASC, for the treatment of complex perianal fistulas in participants with Crohn's disease.

The study will randomize approximately 554 participants.

* Cx601 eASCs intralesional injection
* Placebo - Cx601 placebo-matching eASCs intralesional injection

Study treatments will be allocated, on a 1:1 ratio, by central randomization through interactive web response system (IWRS). The study will follow an add-on design, participants receiving any ongoing concomitant medical treatment, at stable doses at the time of screening, for the CD will be allowed to continue it throughout the study.

The primary efficacy analysis, will be conducted at Week 24 timepoint. The double blind design will be maintained up to Week 52 (both participant and investigator) by a specific blinding for study treatment administration and for evaluating its efficacy.

This multicenter trial will be conducted globally across 150 centers. The overall time to participate in this study is approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Participants of either gender greater than or equal to (>=) 18 years and less than or equal to (<=) 75 years of age.
3. Participants with CD diagnosed at least 6 months prior to Screening visit in accordance with accepted clinical, endoscopic, histological and/or radiological criteria.
4. Presence of complex perianal fistula(s) with a maximum of 2 internal openings and a maximum of 3 external openings based on clinical assessment; a central reading of a locally performed contrast enhanced (gadolinium) pelvic MRI will be performed to confirm location of the fistula and potential associated perianal abscess(es). Fistula(s) must have been draining for at least 6 weeks prior to Screening visit. Actively draining simple subcutaneous fistula(s), at the time of Screening visit, are not allowed in this study. A complex perianal fistula is defined as a fistula that meets one or more of the following criteria :

   * High inter-sphincteric, high trans-sphincteric, extra-sphincteric or suprasphincteric.
   * Presence of >=2 external openings.
   * Associated perianal abscess(es). Note: Abscesses that are larger than 2 cm at least 2 dimensions on MRI must be confirmed to have been drained adequately by the surgeon during the preparation curettage in order to be eligible.
5. Clinically controlled, nonactive or mildly active CD, during the last six months prior to Screening visit with:

   * A patient reported outcomes (PRO-2) score <14 at Screening, AND
   * A colonoscopy documenting the absence of ulcers larger than 0.5 cm in the colonic mucosa:

     - If colonoscopy data are not available within 6 months prior to Screening:
   * A simple endoscopic score for Crohn's Disease (SES-CD) <=6 with absence of rectal ulcers larger than 0.5 cm must be documented in a colonoscopy performed at Screening before randomization.

     - If colonoscopy data are available within 6 months prior to Screening, the following must be documented, otherwise a new colonoscopy (as above) will be mandatory:
   * The absence of ulcers larger than 0.5 cm in the colonic mucosa AND
   * the improvement or no worsening in abdominal pain and/or in the diarrhea, sustained for one week or more, since the last colonoscopy was performed in the clinical records until Screening visit.

   AND

   o No hemoglobin decrease >=2.0 gram per deciliter (g/dL) or an unexplained rising C-reactive protein (CRP), > 5.0 milligram per liter (mg/L) to a concentration above the referenced upper limit of normal (ULN) (unless the rise is due to a known process other than luminal Crohn's Disease), since the last colonoscopy was performed as compared to results during the Screening visit.

   AND

   o no initiation or intensification of treatment with corticosteroids, immunosuppressants or monoclonal antibodies (mAbs) dose regimen since the last endoscopy up to Screening visit.
6. Participants whose perianal fistulas were previously treated and have shown an inadequate response or a loss of response while they were receiving either an immunosuppressive agent or tumour necrosis factor (TNF)-alpha antagonist or vedolizumab or ustekinumab, or having documented intolerance to any of these treatments administered at least at approved or recommended doses during the minimum period mentioned:

   * Immunosuppressive agents: at least 3 months treatment with azathioprine (2-3 milligram per kilogram per day [mg/kg/day]), 6-mercaptopurine (1-1.5 mg/kg/day), or subcutaneous/intramuscular methotrexate (25 mg/week) prior to Screening for the study.
   * TNFalpha antagonists:
   * Infliximab: at least 14 weeks treatment at the approved doses for induction and/or maintenance in Crohn´s disease prior to screening for the study. For induction: 1 intravenous dose of 5 milligram per kilogram (mg/kg) followed by the same dose 2 and 6 weeks after. For maintenance: 5-10 mg/kg intravenously every 8 weeks, or more frequently.
   * Adalimumab: at least 14 weeks treatment at the approved doses for induction and/or maintenance in Crohn's disease prior to screening for the study. For induction: 1 subcutaneous dose of 160 milligram (mg), followed by 80 mg 2 weeks after. For maintenance: 40 mg subcutaneously every other week, or weekly.
   * Certolizumab l: at least 14 weeks treatment at the approved doses for induction and/or maintenance in Crohn´s disease prior to screening for the study. For induction: 1 subcutaneous dose of 400 mg, followed by the same dose 2 and 4 weeks after. For maintenance: 400 mg subcutaneously every 2 to 4 weeks.
   * Anti-integrin: at least 14 weeks treatment of the approved dose for induction and/or maintenance in Crohn´s disease prior to screening for the study. For induction: Vedolizumab 300 mg. For maintenance: Vedolizumab 300 mg every 4 to 8 weeks.
   * Anti-interleukin (IL)-12/23: at least 16 weeks treatment of the approved dose in Crohn´s disease prior to screening for the study. For induction: Ustekinumab, approximately 6mg/kg intravenously initially then followed by 90 mg subcutaneously every 8 weeks.
7. Women of childbearing potential (WCBP) must have negative serum pregnancy test at screening (sensitive to 25 international units [IU] human chorionic gonadotropin [hCG]). Both WCBP or male participants participating in this study, with a WCBP as partner, must agree to use an adequate method of contraception during the entire duration of the study. An adequate method of contraception is defined as complete, non-periodic sexual abstinence (refraining from heterosexual intercourse), single-barrier method, vasectomy, adequate hormonal contraception (to have started at least 7 days prior to Screening visit), or an intra-uterine device (to have been in place for at least 2 months prior to Screening visit).

Exclusion Criteria:

1. Concomitant rectovaginal or rectovesical fistula(s).
2. Participant naïve to prior specific medical treatment for complex perianal fistula(s) including immunosuppressant (IS) or anti-TNFs.
3. Presence of a perianal collection >2 cm in at least two dimensions on the central reading MRI at Screening visit that was not adequately drained as confirmed by the surgeon during the preparation procedure (week -3 to day 0).
4. Severe rectal and/or anal stenosis and/or severe proctitis (defined as the presence of large >0.5 cm ulcers in the rectum) that make impossible to follow the surgery procedure manual.
5. Participant with diverting stomas.
6. Active, uncontrolled infection requiring parenteral antibiotics.
7. Participant with ongoing systemic or rectal steroids for CD in the last 2 weeks prior to the Preparation visit.
8. Participants with major alteration on any of the following laboratory tests or increased risk for the surgical procedure:

   * Serum creatinine levels >1.5 times the ULN
   * Total bilirubin >1.5 ULN
   * Aspartate Transaminase (AST)/ Alanine Transaminase (ALT) >3 times ULN
   * Hemoglobin <10.0 g/dL
   * Platelets <75.0*10^9/L
   * Albuminemia <3.0 g/dL
9. Suspected or documented infectious enterocolitis within two weeks prior to Screening visit.
10. Any prior invasive malignancy diagnosed within the last 5 years prior to Screening visit. Participants with basal-cell carcinoma of the skin completely resected outside the perineal region can be included.
11. Current or recent (within 6 months prior to the Screening visit) history of severe, progressive, and/or uncontrolled hepatic, haematological, gastrointestinal (GI) (other than CD), renal, endocrine, pulmonary, cardiac, neurological or psychiatric disease that may result in participants increased risk from study participation and/or lack of compliance with study procedures.
12. Participants with primary sclerosing cholangitis.
13. Participants with known chronically active hepatopathy of any origin, including cirrhosis and participants with persistent positive Hepatitis B Virus (HBV) surface antigen (HBsAg) and quantitative HBV polymerase chain reaction (PCR), or positive serology for Hepatitis C Virus (HCV) and quantitative HCV PCR within 6 months prior to Screening.
14. Congenital or acquired immunodeficiencies, including participants known to be HIV carriers
15. Known allergies or hypersensitivity to penicillin or aminoglycosides; Dulbecco Modified Eagle's Medium (DMEM); bovine serum; local anaesthetics or gadolinium (MRI contrast).
16. Contraindication to MRI scan (example, due to the presence of pacemakers, hip replacements or severe claustrophobia).
17. Severe trauma within 6 months prior to Screening visit.
18. Pregnant or breastfeeding women.
19. Participants who do not wish to or cannot comply with study procedures.
20. Participants currently receiving, or having received any investigational drug within 3 months prior to Screening visit.
21. Participants previously treated with Cx601 or other allogeneic stem-cell therapy cannot be enrolled into this clinical study.
22. Any major surgery of the GI tract (including one or more segments of the colon or terminal ileum) within 6 months prior the screening or any minor surgery of the GI tract within 3 months prior to screening.
23. Participants who had local perianal surgery other than drainage for the fistula within 6 months prior to the Screening visit, or those who may need surgery in the perianal region for reasons other than fistulas at the time of inclusion in the study.
24. Contraindication to the anaesthetic procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (159):
- United States (68):
  - Scottsdale Mayo Clinic, Scottsdale, Arizona
  - UC San Diego Health Systems, La Jolla, California
  - University of Southern California (USC) Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Medical Center - Chao Family Comprehensive Cancer, Orange, California
  - Inland Empire Liver Foundation, Rialto, California
  - Kaiser Permamente, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Vallejo Hospital and Medical Offices, Vallejo, California
  - Cedar-Sinai Medical Center, West Hollywood, California
  - University of Colorado Hospital, Aurora, Colorado
  - Hartford Hospital - Gastroenterology, Farmington, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic - Gastroenterology, Jacksonville, Florida
  - University of Miami Hospital, Miami, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - USF Health South Tampa Center for Advanced Healthcare, Tampa, Florida
  - Florida Hospital Tampa, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - The University of Chicago Medicine - Colon & Rectal Surgery, Chicago, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Indiana University - Colon and Rectal, Indianapolis, Indiana
  - University of Kansas Sxchool of Medicine, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Digestive Health Center of Louisiana, Baton Rouge, Louisiana
  - Colon and Rectal Surgery Associates, Metairie, Louisiana
  - University Medical Center - New Orleans, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins Medicine - The Johns Hopkins Hospital, Baltimore, Maryland
  - Massachussetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - University of Massachusetts - colon & rectal surgery, Worcester, Massachusetts
  - Mayo Clinic College of Medicine - Division of Colon and Rectal Surgery - Division of Colon and Rectal Surgery, Rochester, Minnesota
  - Barnes-Jewish Hospital - Gastroenterology, St Louis, Missouri
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center - Cancer Center, Lebanon, New Hampshire
  - Morristown Medical Center - Gastroenterology, Morristown, New Jersey
  - Albany Medical Center, Albany, New York
  - North Shore University Hospital - Gastroenterology, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - Stony Brook University Medical Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - OHSU Digestive Health Center, Portland, Oregon
  - Harvard Medical School-Beth Israel Deaconess Medical Center, Hershey, Pennsylvania
  - Penn State Hershey Medical Center - Surgery, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University Surgical Associates-Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Rapid City Medical Center, Rapid City, South Dakota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center - Gastroenterology - Gastroenterology, Dallas, Texas
  - Baylor College of Medicine (BCM) - Gastroenterology, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - Virginia Mason Medical Center - Gastroenterology, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Hub for Collaborative Medicine - Gastroenterology and Hepatology, Milwaukee, Wisconsin
- Belgium (9):
  - UZ Leuven - Campus Gasthuisberg, Leuven, Vlaams Brabant
  - AZ Groeninge - Campus Kennedylaan - Gastro-enterology, Kortrijk, West-Vlaanderen
  - AZ Delta vzw - Maag-darm-leverziekten, Roeselare, West-Vlaanderen
  - GZA ziekenhuizen - Campus Sint-Vincentius - Gastro-enterology, Antwerp
  - Imelda Ziekenhuis, Antwerp
  - UZ Gent - Gastroenterology, Ghent
  - CHU de Liege - Domaine Universitaire du Sart Tilman, Liège
  - Clinique Saint-Joseph (CHC), Liège
  - CHU Dinant Godinne UCL Namur, Namur
- Canada (7):
  - University of Alberta, Edmonton, Alberta
  - (G.I.R.I.) GI Research Institute, Vancouver, British Columbia
  - Ottawa Hospital, Ottawa, Ontario
  - Mount Sinai Hospital - Toronto - Gastroenterology, Toronto, Ontario
  - Kensington Screening Clinic - Gastroenterology, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University Health Centre - Montreal General Hospital, Montreal, Quebec
- Czechia (2):
  - NH Hospital a.s., Hořovice, Beroun
  - FN Hradec Kralove, Hradec Králové
- Denmark (3):
  - Bispebjerg Hospital, Copenhagen, Copenhague
  - Aarhus University Hospital - Department of Hepatology and Gastroenterology, Lever-Mave- og Tarmsygdomme Klinik, krydspunkt C216, Aarhus
  - Odense Universitetshospital, Odense
- France (12):
  - CHU de Nice, Nice, Alpes-Maritimes
  - CHU de Clermont-Ferrand - Estaing, Clermont-Ferrand, Auvergne
  - Centre Hospitalier Universitaire De Toulouse - Hopital De Ra, Toulouse, Haute-Garonne
  - CHRU Hopital De Pontchaillou, Rennes, Ille-et-Vilaine
  - CHRU de Nancy -Hopital Brabois Adultes - Service d'Hepato- Gastroenterologie, Vandœuvre-lès-Nancy, Lorraine
  - CHRU De Lille - Hopital Claude Huriez - Hepato-Gastro-Enterologie, Lille, Nord
  - CHU Saint Etienne, Saint Priest En Jarez, Pays de la Loire Region
  - CHU Amiens-Picardie, Amiens, Picardie
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhone
  - Paris St. Joseph Hospital, Paris
  - Hopital Beaujon, Clichy, Île-de-France Region
  - Hopital Saint Louis - Gastro-hepatoenterologie, Paris, Île-de-France Region
- Germany (4):
  - Universitatsklinikum Erlangen, Erlangen, Bavaria
  - Klinikum der Universitat Munchen - Campus Grosshadern, München, Bavaria
  - Klinikum der Johann Wolfgang Goethe-Universitat, Frankfurt am Main, Hesse
  - Universitatsklinikum Dresden, Dresden, Saxony
- Hungary (4):
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont - I. sz. Belgyogyaszati Klinika, Szeged, Csongrád megye
  - Debreceni Egyetem Klinikai Kozpont, Debrecen, Hajdú-Bihar
  - MH Egeszsegugyi Kozpont - Gasztroenterologiai Osztaly, Budapest, Pest County
  - Semmelweis Egyetem, Budapest, Pest County
- Israel (5):
  - Rabin Med Ctr Beilinson Hosp, Petah Tikva, Central District
  - Shaare Zedek Medical Center - Gastroenterology, Jerusalem, Jerusalem
  - Hadassah Medical Organization, Hadassah Medical Center, Ein-, Jerusalem, Jerusalem
  - Rambam Medical Centre, Haifa, Northern District
  - Chaim sheba Medical Center, Tel Litwinsky, Tel Aviv
- Italy (13):
  - Ospedale Santissima Annunziata, Cento, Ferrara
  - Istituto Clinico Humanitas Rozzano, IRCCS - IBD Center, Rozzano, Milano
  - Policlinico S. Orsola Malpighi, AOU di Bologna-U.O. di Medicina Interna., Bologna
  - AOU Policlinico di Modena - Gastroenterologia, Modena
  - II Universita degli Studi di Napoli, Napoli
  - Gastroenterology Section, Palermo
  - Universita degli studi di Pisa, Pisa
  - Policlinico Universitario Campus Biomedico - UOC di Gastroenterologia, Roma
  - A.O. San Camillo Forlanini, Roma
  - Complesso Integrato Columbus, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliero Universitaria S.Maria della Misericordia - Gastroenterologia, Udine
  - Azienda Ospedaliera Universitaria Integrata Verona (AOUI) -, Verona
- Poland (7):
  - Centrum Medyczne PROMED, Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne Melita Medical, Wroclaw, Lower Silesian Voivodeship
  - Wielospecjalistyczny Szpital Medicover, Warsaw, Masovian Voivodeship
  - Endoskopia Sp z o.o., Sopot, Pomeranian Voivodeship
  - COPERNICUS Podmiot Leczniczy Sp. z o.o., Gdansk
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Wojskowej Akademii Medycznej Centralny Szpital Weteranow, Lodz, Łódź Voivodeship
- University of Puerto Rico School of Medicine, San Juan, Puerto Rico
- Spain (15):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - H.U. G.Trias i Pujol, Badalona, Barcelona
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital de Sagunto, Sagunto, Valencia
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - C.H.U. de Pontevedra, Pontevedra
  - H.U.V. del Rocio, Seville
- Linkoping University Hospital - Department of Surgery, Linköping, Ostergotlands Lan [se-05], Sweden
- United Kingdom (8):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - NHS Greater Glasgow and Clyde - Glasgow Royal Infirmary (GRI), Glasgow, Glasgow City
  - St. Mark's Hospital, Harrow, London, City of
  - Guys & St Thomas, London, London, City of
  - Nottingham University Hospitals NHS Trust - Surgery, Nottingham, Nottinghamshire
  - University Colleague London Hospital (UCLH), London
  - Wythenshawe Hospital - Gastroenterology, Manchester
  - Northern General Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 113 investigative sites in Belgium, Czechia, Denmark, France, Germany, Hungary, Israel, Italy, Poland, Spain, United Kingdom, Canada, and United States from 15 September 2017 to 26 July 2023.
Pre-assignment Details: A total of 568 participants with a diagnosis of Crohn's disease were enrolled in a 1:1 ratio to receive either Cx601 or matching placebo.
Period: Overall Study
Arm/Group | Placebo | Cx601
Started | 285 | 283
Completed | 246 | 249
Not Completed | 39 | 34
Not completed — Withdrawal by Subject | 12 | 20
Not completed — Physician Decision | 4 | 1
Not completed — Lost to Follow-up | 8 | 8
Not completed — Death | 0 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Reason not Specified | 14 | 4

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) Analysis Set included all randomized participants regardless of their being treated or not and regardless of their having any postbaseline efficacy measurements or not.
Groups:
- Placebo: Placebo (saline) 24 mL was administered once by local injection.
- Cx601: Cx601 eASCs 120 million cells (5 million cells/mL) was administered once by local injection.
- Total: Total of all reporting groups
Arm/Group | Placebo | Cx601 | Total
Number analyzed (Participants) | 285 | 283 | 568
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (10.78) | 38.4 (11.91) | 38.1 (11.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 121 | 251
  Male | 155 | 162 | 317
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 13 | 26
  Not Hispanic or Latino | 250 | 240 | 490
  Unknown or Not Reported | 22 | 30 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 8 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 254 | 243 | 497
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 18 | 24 | 42
Height [Mean (Standard Deviation); unit: centimeters (cm)] — Population: Number of participants analyzed is the number of participants with data available for height at the Baseline.
  centimeters (cm)
    number analyzed (Participants) | 274 | 278 | 552
    (all) | 171.78 (9.088) | 171.59 (9.429) | 171.69 (9.253)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] — Population: Number of participants analyzed is the number of participants with data available for weight at the Baseline.
  kilograms (kg)
    number analyzed (Participants) | 274 | 278 | 552
    (all) | 77.69 (16.675) | 78.73 (19.620) | 78.21 (18.209)
Body Mass Index (BMI) [Count of Participants; unit: Participants] — Population: Number of participants analyzed is the number of participants with data available for BMI at the Baseline.
  Participants
    number analyzed (Participants) | 274 | 278 | 552
    Less than 18.5 kilograms per square meter(kg/m^2) | 4 | 9 | 13
    18.5 to <25.0 kg/m^2 | 132 | 110 | 242
    25.0 to <30.0 kg/m^2 | 81 | 92 | 173
    30.0 kg/m^2 or Higher | 57 | 67 | 124

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Combined Remission at Week 24
Description: Combined remission was defined as the closure of all treated external openings that were draining at baseline despite gentle finger compression and absence of collection(s) >2 cm (in at least 2 dimensions) of the treated perianal fistula(s) confirmed by blinded central magnetic resonance imaging (MRI) assessment. Percentages are rounded off to whole number at the nearest decimal.
Time Frame: Week 24
Population: The ITT Analysis Set included all randomized participants regardless of their being treated or not and regardless of their having any postbaseline efficacy measurements or not.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cx601
Number analyzed (Participants) | 285 | 283
percentage of participants | 46.32 [40.53 to 52.10] | 48.76 [42.94 to 54.59]
Statistical Analysis 1: Comparison: Placebo vs Cx601; Test type: Superiority; p = 0.571, Cochran-Mantel-Haenszel — P-value was based on stratified Cochran-Mantel-Haenszel (CMH) test adjusting for interactive web response system (IWRS) randomization stratification factors; Difference in Combined Remission Rate = 2.37, 95% CI 2-sided [-5.82 to 10.55] — The asymptotic Wald's confidence intervals (CI) are displayed

2. Secondary Outcome: Percentage of Participants With Clinical Remission at Week 24
Description: Clinical remission was defined as closure of all treated external openings that were draining at baseline despite gentle finger compression. Percentages are rounded off to whole number at the nearest decimal.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cx601
Number analyzed (Participants) | 285 | 283
percentage of participants | 47.02 [41.22 to 52.81] | 49.82 [44.00 to 55.65]
Statistical Analysis 1: Comparison: Placebo vs Cx601; Test type: Superiority; p = 0.515, Cochran-Mantel-Haenszel — P-value was based on stratified CMH test adjusting for IWRS randomization stratification factors; Difference in Clinical Remission Rate = 2.72, 95% CI 2-sided [-5.47 to 10.90] — The asymptotic Wald's confidence intervals are displayed

3. Secondary Outcome: Time to Clinical Remission at Week 24
Description: Time to clinical remission was defined as the time from treatment start to first visit with closure of all treated external openings that were draining at baseline despite gentle finger compression, as clinically assessed.
Time Frame: Week 24
Population: The ITT Analysis Set included all randomized participants regardless of their being treated or not and regardless of their having any postbaseline efficacy measurements or not. Overall number analyzed is the number of participants who had clinical remission at Week 24.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Cx601
Number analyzed (Participants) | 134 | 141
weeks | 7.14 [7.00 to 11.29] | 7.00 [6.71 to 7.29]
Statistical Analysis 1: Comparison: Placebo vs Cx601; Test type: Superiority; p = 0.374, Log Rank — P-value was based on a stratified log-rank test adjusting for IWRS randomization stratification factors; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.90 to 1.32] — Cox Proportional Hazard Regression model was used to estimate the hazard ratio and 95% CI, adjusting for IWRS randomization stratification factors

4. Secondary Outcome: Percentage of Participants With Combined Remission at Week 52
Description: Combined remission was defined as the closure of all treated external openings that were draining at baseline despite gentle finger compression, and absence of collections >2 cm (in at least 2 dimensions) confirmed by blinded central MRI assessment. Percentages are rounded off to whole number at the nearest decimal.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cx601
Number analyzed (Participants) | 285 | 283
percentage of participants | 39.65 [33.97 to 45.33] | 40.99 [35.26 to 46.72]
Statistical Analysis 1: Comparison: Placebo vs Cx601; Test type: Superiority; p = 0.757, Cochran-Mantel-Haenszel — P-value was based on stratified CMH test adjusting for IWRS randomization stratification factors; Difference in Combined Remission Rate = 1.27, 95% CI 2-sided [-6.77 to 9.31] — The asymptotic Wald's confidence intervals are displayed

5. Secondary Outcome: Percentage of Participants With Clinical Remission at Week 52
Description: as for outcome 2
Time Frame: Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cx601
Number analyzed (Participants) | 285 | 283
percentage of participants | 41.40 [35.69 to 47.12] | 43.11 [37.34 to 48.88]
Statistical Analysis 1: Comparison: Placebo vs Cx601; Test type: Superiority; p = 0.697, Cochran-Mantel-Haenszel — P-value was based on stratified CMH test adjusting for IWRS randomization stratification factors; Difference in Clinical Remission Rate = 1.60, 95% CI 2-sided [-6.46 to 9.66] — The asymptotic Wald's confidence intervals are displayed

6. Secondary Outcome: Percentage of Participants With Clinical Response at Week 24
Description: Clinical response was defined as closure of at least 50 percent (%) of all treated external openings that were draining at baseline despite gentle finger compression. Percentages are rounded off to whole number at the nearest decimal.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cx601
Number analyzed (Participants) | 285 | 283
percentage of participants | 58.60 [52.88 to 64.31] | 61.84 [56.18 to 67.50]
Statistical Analysis 1: Comparison: Placebo vs Cx601; Test type: Superiority; p = 0.428, Cochran-Mantel-Haenszel — P-value was based on stratified CMH test adjusting for IWRS randomization stratification factors; Difference in Clinical Response Rate = 3.23, 95% CI 2-sided [-4.76 to 11.21] — The asymptotic Wald's confidence intervals are displayed

7. Secondary Outcome: Percentage of Participants With Clinical Response at Week 52
Description: Clinical response was defined as closure of at least 50% of all treated external openings that were draining at baseline, despite gentle finger compression. Percentages are rounded off to whole number at the nearest decimal.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cx601
Number analyzed (Participants) | 285 | 283
percentage of participants | 50.88 [45.07 to 56.68] | 53.71 [47.90 to 59.52]
Statistical Analysis 1: Comparison: Placebo vs Cx601; Test type: Superiority; p = 0.497, Cochran-Mantel-Haenszel — P-value was based on stratified CMH test adjusting for IWRS randomization stratification factors; Difference in Clinical Response Rate = 2.84, 95% CI 2-sided [-5.35 to 11.03] — The asymptotic Wald's confidence intervals are displayed

8. Secondary Outcome: Time to Clinical Remission at Week 52
Description: as for outcome 3
Time Frame: Week 52
Population: The ITT Analysis Set included all randomized participants regardless of their being treated or not and regardless of their having any postbaseline efficacy measurements or not. Overall number analyzed is the number of participants with clinical remission at Week 52.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Cx601
Number analyzed (Participants) | 118 | 122
weeks | 7.14 [7.00 to 11.29] | 7.00 [6.71 to 7.29]
Statistical Analysis 1: Comparison: Placebo vs Cx601; Test type: Superiority; p = 0.363, Log Rank — P-value was based on a stratified log-rank test adjusting for IWRS randomization stratification factors; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.90 to 1.32] — Cox Proportional Hazard Regression model was used to estimate hazard ratio and 95% CI, adjusting for IWRS randomization stratification factors

9. Secondary Outcome: Time to Clinical Response at Week 24
Description: Time to clinical response was defined as the time from treatment start to first visit with closure of at least 50% of all treated external openings that were draining at baseline, despite gentle finger compression, as clinically assessed.
Time Frame: Week 24
Population: The ITT Analysis Set included all randomized participants regardless of their being treated or not and regardless of their having any postbaseline efficacy measurements or not. Overall number analyzed is the number of participants with clinical response at Week 24.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Cx601
Number analyzed (Participants) | 167 | 175
weeks | 6.71 [6.29 to 6.86] | 6.71 [6.43 to 7.00]
Statistical Analysis 1: Comparison: Placebo vs Cx601; Test type: Superiority; p = 0.833, Log Rank — P-value was based on a stratified log-rank test adjusting for IWRS randomization stratification factors; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.82 to 1.18] — [estimate comment as in outcome 8, analysis 1]

10. Secondary Outcome: Time to Clinical Response at Week 52
Description: Time to clinical response was defined as time from treatment start to first visit with closure of at least 50% of all treated external openings that were draining at baseline despite gentle finger compression, as clinically assessed.
Time Frame: Week 52
Population: The ITT Analysis Set included all randomized participants regardless of their being treated or not and regardless of their having any postbaseline efficacy measurements or not. Overall number analyzed is the number of participants with clinical response at Week 52.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Cx601
Number analyzed (Participants) | 145 | 152
weeks | 6.71 [6.29 to 6.86] | 6.71 [6.43 to 7.00]
Statistical Analysis 1: Comparison: Placebo vs Cx601; Test type: Superiority; p = 0.717, Log Rank — P-value was based on a stratified log-rank test adjusting for IWRS randomization stratification factors; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.81 to 1.16] — [estimate comment as in outcome 8, analysis 1]

11. Secondary Outcome: Percentage of Participants With Relapse by Week 52 After Achieving Combined Remission at Week 24
Description: Relapse was defined as reopening of any of the treated fistulas external openings with active drainage as clinically assessed, or the development of a perianal fluid collection >2 cm of the treated perianal fistula confirmed by centrally read MRI assessment in participants who were in combined remission at week 24. Percentages are rounded off to whole number at the nearest decimal.
Time Frame: From Week 24 to Week 52
Population: The ITT Analysis Set included all randomized participants regardless of their being treated or not and regardless of their having any postbaseline efficacy measurements or not. Overall number analyzed is the number of participants who were responders (achieved combined remission) at Week 24.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cx601
Number analyzed (Participants) | 132 | 138
percentage of participants | 31.06 [23.17 to 38.95] | 34.06 [26.15 to 41.96]
Statistical Analysis 1: Comparison: Placebo vs Cx601; Test type: Superiority; p = 0.599, Cochran-Mantel-Haenszel — P-value was based on stratified CMH test adjusting for IWRS randomization stratification factors; Difference in Relapse Rate = 3.03, 95% CI 2-sided [-8.28 to 14.34] — The asymptotic Wald's confidence intervals are displayed

12. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Treatment-emergent Serious Adverse Events (TESAEs), and Treatment-emergent Adverse Events of Special Interest (TEAESIs)
Description: An adverse event(AE)=any untoward medical occurrence in a clinical investigation participant receiving a medicinal product; it did not necessarily have to have a causal relationship with this treatment. Serious adverse event(SAE)=any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization/prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or was a congenital abnormality/birth defect, or was a medically significant event or required intervention to prevent at least one of the outcomes listed above, or was a suspected transmission of an infectious agent. AESIs included tumorigenicity, ectopic tissue formation, hypersensitivity reactions, transmission of infectious agents, immunogenicity/alloimmune reactions, and medication errors, as reported by the investigator. TEAE=AE whose onset occurred, severity worsened, or intensity increased after receiving the study treatment.
Time Frame: From first dose of study drug to end of follow up period (up to Week 52)
Population: The Safety (SAF) Analysis Set included all randomized participants who received the actual study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cx601
Number analyzed (Participants) | 274 | 278
Participants
  TEAEs | 201 | 203
  TESAEs | 35 | 41
  TEAESIs | 3 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Sign Parameters
Description: Vital signs included measurement of pulse rate, systolic and diastolic blood pressure, respiratory rate, and body temperature. Clinically significant vital signs assessment was based on investigator interpretation. Number of participants with clinically significant changes in vital signs were reported.
Time Frame: From first dose of study drug to end of follow up period (up to Week 52)
Population: SAF Analysis Set included all randomized participants who received the actual study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cx601
Number analyzed (Participants) | 274 | 278
Participants | 0 | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Parameters
Description: Laboratory parameters included blood chemistry and hematology. Clinically significant laboratory parameters assessment was based on investigator interpretation. Number of participants with clinically significant changes in laboratory parameters (hematology and blood chemistry) were reported.
Time Frame: From first dose of study drug to end of follow up period (up to Week 52)
Population: SAF Analysis Set included all randomized participants who received the actual study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cx601
Number analyzed (Participants) | 274 | 278
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug to end of follow up period (up to Week 52)
Description: All-cause Mortality: ITT Analysis Set included all randomized participants regardless of their being treated or not and regardless of their having any postbaseline efficacy measurements or not. Serious and Other Adverse Events: SAF Analysis Set included all randomized participants who received the actual study treatment.
Arm/Group | Placebo | Cx601
All-Cause Mortality (participants affected / at risk) | 0/285 | 1/283
Serious Adverse Events (participants affected / at risk) | 35/274 | 41/278
Other Adverse Events (participants affected / at risk) | 67/274 | 66/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=274) | Cx601 (N=278)
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abscess limb (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 12 | 12
Anal fistula (Gastrointestinal disorders) | 4 | 4
Anal inflammation (Gastrointestinal disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0
Anorectal disorder (Gastrointestinal disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 3
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 2 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/130 | 0/121 — Number of participants at risk in each arm is based on the female population in this study.
Female genital tract fistula (Reproductive system and breast disorders) | 1/130 | 1/121 — Number of participants at risk in each arm is based on the female population in this study.
Gastroenteritis (Infections and infestations) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Histoplasmosis disseminated (Infections and infestations) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/130 | 0/121 — Number of participants at risk in each arm is based on the female population in this study.
Perirectal abscess (Infections and infestations) | 1 | 1
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Subileus (Gastrointestinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=274) | Cx601 (N=278)
COVID-19 (Infections and infestations) | 22 | 21
Crohn's disease (Gastrointestinal disorders) | 16 | 13
Proctalgia (Gastrointestinal disorders) | 40 | 40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi-site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/81/NCT03279081/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT03279081/SAP_001.pdf